CLINICAL TRIAL: NCT01265537
Title: A Prospective, Open Label, Pilot Study Comparing the Use of Low-target Advagraf With Rabbit Antithymocyte Globulin Induction Versus Conventional Target Advagraf With Basiliximab Induction in a Steroid-avoidance Immunosuppressive Protocol for de Novo Renal Transplant Recipients
Brief Title: A Pilot Study Comparing the Use of Low-target Versus Conventional Target Advagraf
Acronym: Astellas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Astellas Pharma Canada, Inc. (Industry)
Responsible Party: Principal Investigator, Jagbir Gill, Assistant Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H10-03047
Record Dates: First submitted 2010-12-21; First posted 2010-12-23 (Estimated); Results first posted 2020-02-11 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Acute Graft Rejection; Diabetes
Keywords: Transplant; Tacrolimus; Diabetes after transplant; Acute rejection prevention; New onset diabetes after transplant
MeSH Terms: conditions — Diabetes Mellitus | interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low target tacrolimus (Advagraf) (Experimental): This group will receive rabbit anti-thymocyte globulin (rATG) induction (3 -4 doses of 1.5 mg/kg during the first post transplant week) with IV solumedrol, MPA (Mycophenolate Mofetil or Mycophenolate Sodium), and "low-target" Advagraf.
  Interventions: Drug: Tacrolimus
- Standard target tacrolimus (Advagraf) (Active Comparator): This group will receive basiliximab induction (40 mg total) with IV solumedrol, MPA (Mycophenolate Mofetil or Mycophenolate Sodium), and "standard target" Advagraf.
  Interventions: Drug: Tacrolimus

INTERVENTIONS:
Drug: Tacrolimus — Low target tacrolimus Advagraf (0.25mg/kg) orally once daily dosed as per manufacturer's recommendation to target trough levels as per Table 1
  Table 1
  Months post tx:
  0-1 month, level 5-7; 1-3 months, level 4-5; and 3-6 months, level 3-4
  Other Names: Advagraf
  Arms: Low target tacrolimus (Advagraf)
Drug: Tacrolimus — Standard dose of tacrolimus Advagraf (0.25mg/kg) orally once daily dosed as per manufacturer's recommendation to target trough levels as per Table 1
  Table 1
  Months post tx
  0-1 month; level 8-12; 1-3 months, level 6-9; and 3-6 months, level 5-8.
  Other Names: Advagraf
  Arms: Standard target tacrolimus (Advagraf)

SUMMARY:
While the incidence of acute rejection and early graft loss have improved dramatically with the advent of newer immunosuppressant medications, improvements in long-term patient and allograft survival after kidney transplantation have not been achieved. The specific drug combination that provides the best outcomes with the least amount of side effects is not known. Each kidney transplant center uses the combination of drugs that they believe is optimal. This study is about identifying whether drugs that are currently approved for use in kidney transplantation can be used in a new combination safely and with potentially fewer side effects than the drug combinations that are currently used at St. Paul's Hospital and other transplant centres.

DETAILED DESCRIPTION:
Purpose This study has been designed to test whether using Thymoglobulin with low dose tacrolimus and early steroid withdrawal will minimize both kidney rejection and the development of new onset diabetes after transplant (NODAT).

Justification Experimental treatment is low target tacrolimus with thymoglobulin. Standard treatment is a standard target (higher dose) tacrolimus and basiliximab, instead of thymoglobulin.

The investigators hypothesize, that a combined approach of early steroid withdrawal and low dose tacrolimus in low immunologic risk transplant recipients will be effective in reducing the incidence of new onset diabetes mellitus, while maintaining a low risk of acute rejection.

Objective

The objective of this study is to compare early post-transplant outcomes with the use of low target versus standard target Advagraf in de novo kidney allograft recipients of low immunologic risk undergoing early corticosteroid withdrawal.

Research Method

This is a pilot study. Primary and secondary outcomes are as follows:

Primary Outcome Composite endpoint of biopsy proven acute rejection and NODAT at 6 months post transplantation.

Secondary Outcomes

* Patient survival
* Graft survival
* Frequency, severity, and treatment of hypertension
* Frequency, severity, and treatment of hyperlipidemia (serum total cholesterol, (high density lipoprotein (HDL), low-density lipoprotein (LDL), and triglycerides)
* Weight gain
* Infections (cytomegalovirus (CMV), opportunistic infections including urinary tract infections requiring treatment, pneumonia)
* Malignancy, including post-transplant lymphoproliferative disease (PTLD)
* Leukopenia
* Renal function as measured by serum creatinine and estimated Glomerular Filtration Rate (eGFR)

The primary endpoint will be evaluated by time-to-event Kaplan Meier analysis and by Chi-squared analysis of final 6 month data.

Statistical Analysis

Sample size and power:

In the setting of early steroid withdrawal, Woodle et al. reported an acute rejection rate of 14% with rATG and 24% with an interleukin-2 receptor antibody induction(10). The incidence of NODAT was reported at 21% by Woodle, et al., and was reported 10% in the low dose tacrolimus arm of the ELITE-Symphony trial. The investigators, therefore expect a combined event rate of 24% in Group A and 45% in group B. With a power of 0.80 and alpha error of 0.05, the investigators determined that the investigators need 72 subjects in each arm to demonstrate a 20% difference in our composite primary outcome. For this initial pilot study, the investigators aim to recruit a total of 30 subjects After receiving informed consent, subjects will be randomized on a 1:1 basis to one of the two treatment groups. Subjects who discontinue the study prematurely will not be replaced.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients over 18 years of age who receive a deceased, living unrelated or living related donor renal transplant
2. No history of pre-existing diabetes mellitus
3. Not using diabetic medications (insulin, hypoglycemic agents) at the time of transplantation
4. Random plasma glucose level <11.1 at the time of transplantation
5. Peak PRA (panel reactive antibody) <30%
6. Females capable of becoming pregnant must have a negative pregnancy test at baseline and are required to practice an approved method of birth control for the duration of the study and for a period of three months following discontinuation of study medication
7. The patient has given written informed consent to participate in the study

Exclusion Criteria:

1. Patients with primary non-function
2. Peak PRA>=30%
3. Multiple organ transplants
4. HLA (human leukocyte antigen) identical living donor transplant recipients
5. Cold ischemia time over 36 hours
6. Nonheart beating donor kidney recipients
7. Pediatric donor kidney recipients
8. Donor age>=65 years
9. Patients who are known to have a positive hepatitis C serology, who are human immunodeficiency virus (HIV) or Hepatitis B surface antigen positive. Laboratory results obtained within 6 months prior to study entry are acceptable. Recipients of organs from donors who test positive for Hepatitis B surface antigen or Hepatitis C will be excluded.
10. Patients who are Epstein-Barr virus (EBV) negative and are receiving a transplant from an EBV-positive donor (mismatch).
11. Presence of any severe allergy requiring acute (within 4 weeks of baseline) or chronic treatment, or hypersensitivity to drugs similar to those used in the study
12. Patients with systemic infections
13. Existence of any surgical or medical condition, other than the current transplant, which in the opinion of the investigator, preclude enrollment in this trial
14. Inability to cooperate or communicate with the investigator

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-06-24 (Actual); Primary Completion 2019-02-21 (Actual); Study Completion 2019-10-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jagbir Gill, MD, Principal Investigator — UBC / Dept of Medicine / Nephrology
Locations (1):
- St. Paul's Hospital, Vancouver, British Columbia, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- Low Target Tacrolimus (Advagraf): This group will receive rabbit anti-thymocyte globulin (rATG) induction (3 -4 doses of 1.5 mg/kg during the first post transplant week) with IV solumedrol, MPA (Mycophenolate Mofetil or Mycophenolate Sodium), and "low-target" Advagraf.
  Tacrolimus: Low target tacrolimus Advagraf (0.25mg/kg) orally once daily dosed as per manufacturer's recommendation to target trough levels as per Table 1
  Table 1
  Months post tx:
  0-1 month, level 5-7; 1-3 months, level 4-5; and 3-6 months, level 3-4
- Standard Target Tacrolimus (Advagraf): This group will receive basiliximab induction (40 mg total) with IV solumedrol, MPA (Mycophenolate Mofetil or Mycophenolate Sodium), and "standard target" Advagraf.
  Tacrolimus: Standard dose of tacrolimus Advagraf (0.25mg/kg) orally once daily dosed as per manufacturer's recommendation to target trough levels as per Table 1
  Table 1
  Months post tx
  0-1 month; level 8-12; 1-3 months, level 6-9; and 3-6 months, level 5-8.
Period: Overall Study
Arm/Group | Low Target Tacrolimus (Advagraf) | Standard Target Tacrolimus (Advagraf)
Started | 15 | 15
Completed | 13 | 13
Not Completed | 2 | 2
Not completed — Adverse Event | 2 | 1
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Population: The discrepancy in the Baseline Analysis Population Description and the Overall Number of Baseline Participants is seen because 28 participants in total completed their baseline assessments.
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Target Tacrolimus (Advagraf) | Standard Target Tacrolimus (Advagraf) | Total
Number analyzed (Participants) | 14 | 14 | 28
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 61.8 [49.2 to 66.6] | 50.4 [46.6 to 56.5] | 54.3 [47.1 to 62.7]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 10 | 10 | 20
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 4 | 4
  Caucasian/White | 13 | 9 | 22
  Other/Multiracial | 1 | 0 | 1
  Pacific Islander | 0 | 1 | 1
Family History of Diabetes [Number; unit: participants] | 6 | 6 | 12
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 25.1 (3.0) | 27.5 (6.3) | 26.4 (5.1)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 150 (21) | 159 (27) | 154 (24)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 81 (9) | 87 (9) | 84 (9)
Cholesterol Medications [Count of Participants; unit: Participants]
  Yes | 4 | 2 | 6
  No | 10 | 12 | 22
Cholestoral [Mean (Standard Deviation); unit: mmol/L] | 4.56 (0.97) | 4.43 (0.60) | 4.49 (0.78)
Low-Density Lipoproteins [Mean (Standard Deviation); unit: mmol/L] | 2.72 (0.82) | 2.68 (0.76) | 2.70 (0.77)
High-Density Lipoproteins [Mean (Standard Deviation); unit: mmol/L] | 1.21 (0.28) | 1.37 (0.62) | 1.30 (0.49)
Triglycerides [Mean (Standard Deviation); unit: mmol/L] | 1.38 (0.36) | 1.52 (1.08) | 1.46 (0.82)
Fasting Glucose [Mean (Standard Deviation); unit: mmol/L] | 5.6 (0.8) | 5.2 (0.6) | 5.4 (0.7)
Random Glucose [Mean (Standard Deviation); unit: mmol/L] | 5.5 (1.3) | 5.7 (1.1) | 5.6 (1.2)
Peak Panel-Reactive Antibody (PRA) before transplant [Median (Full Range); unit: %] — Panel reactive antibody (PRA) testing is performed on patients prior to transplantation in an effort to identify the potential presence of anti-HLA antibodies and minimize the risk of antibody mediated rejection. The inclusion criteria for this study was a peak PRA <30%.
  % | 0 [0 to 9] | 0 [0 to 6] | 0 [0 to 9]
Donor Type [Number; unit: participants]
  Living | 11 | 3 | 14
  Deceased | 3 | 11 | 14
Donor Age [Median (Inter-Quartile Range); unit: years] | 41 [33 to 53] | 34 [26 to 56] | 39 [31 to 54]
Human Leukocyte Antigen (HLA) Matches [Count of Participants; unit: Participants] — Human Leukocyte Antigen (HLA) testing is done before an organ transplant to find out if tissues match between the donor and the person receiving the transplant.
  Participants
    0 matches | 3 | 6 | 9
    1 match | 4 | 3 | 7
    2 matches | 3 | 0 | 3
    3 matches | 1 | 1 | 2
    4 matches | 1 | 0 | 1
    5 matches | 1 | 0 | 1
    Missing | 1 | 4 | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With New Onset Diabetes After Transplant (NODAT) or Acute Rejection
Description: Composite endpoint of biopsy proven acute rejection and NODAT at 6 months post transplantation. NODAT will be defined as either FPG >7.0mmol/L OR symptoms of hyperglycemia and a random plasma glucose of >11.1 OR 2-h plasma glucose >11.1 during an oral glucose tolerance test(OGTT).
Time Frame: 6 months post transplant
Population: The discrepancy in the overall number of participants with outcome measure data and the overall number of participants in the participant flow module is seen because 28 participants in total have outcome measure data available.
Measure: Count of Participants; unit: Participants
Arm/Group | Low Target Tacrolimus (Advagraf) | Standard Target Tacrolimus (Advagraf)
Number analyzed (Participants) | 14 | 14
Participants | 2 | 2

2. Secondary Outcome: Number of Participant Deaths
Description: Death of any participant by end of study.
Time Frame: 6 months post transplant
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Low Target Tacrolimus (Advagraf) | Standard Target Tacrolimus (Advagraf)
Number analyzed (Participants) | 14 | 14
Participants | 0 | 0

3. Secondary Outcome: Number of Participants With Graft Failure
Description: Any graft failure by the end of the study.
Time Frame: 6 months post transplant
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Low Target Tacrolimus (Advagraf) | Standard Target Tacrolimus (Advagraf)
Number analyzed (Participants) | 14 | 14
Participants | 0 | 0

4. Secondary Outcome: Number of Participants With Dialysis Events
Description: Any dialysis required by end of study.
Time Frame: 6 months post transplant
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Low Target Tacrolimus (Advagraf) | Standard Target Tacrolimus (Advagraf)
Number analyzed (Participants) | 14 | 14
Participants | 1 | 3

5. Secondary Outcome: Number of Participants With Infection Events
Description: Any infection (CMV, opportunistic infections including urinary tract infections requiring treatment, pneumonia) by end of study.
Time Frame: 6 months post transplant
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Low Target Tacrolimus (Advagraf) | Standard Target Tacrolimus (Advagraf)
Number analyzed (Participants) | 14 | 14
Participants | 5 | 5

6. Secondary Outcome: Number of Participants With Hospitalization Events
Description: Any hospitalization by end of study.
Time Frame: 6 months post transplant
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Low Target Tacrolimus (Advagraf) | Standard Target Tacrolimus (Advagraf)
Number analyzed (Participants) | 14 | 14
Participants | 0 | 4

7. Secondary Outcome: Number of Participants With Malignancy Events
Description: Any malignancy (including post-transplant lymphoproliferative disease) by end of study.
Time Frame: 6 months post transplant
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Low Target Tacrolimus (Advagraf) | Standard Target Tacrolimus (Advagraf)
Number analyzed (Participants) | 14 | 14
Participants | 0 | 1

8. Secondary Outcome: Number of Participants With Cardiovascular Event
Description: Any cardiovascular events by end of study.
Time Frame: 6 months post transplant
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Low Target Tacrolimus (Advagraf) | Standard Target Tacrolimus (Advagraf)
Number analyzed (Participants) | 14 | 14
Participants | 0 | 0

9. Secondary Outcome: Number of Any Leukopenia Events
Description: Any leukopenia by end of study.
Time Frame: 6 months post transplant
Population: as for outcome 1
Measure: Number; unit: events
Arm/Group | Low Target Tacrolimus (Advagraf) | Standard Target Tacrolimus (Advagraf)
Number analyzed (Participants) | 14 | 14
events | 11 | 3

10. Secondary Outcome: Number of Leukopenia Events on ≥2 Occasions
Description: Any leukopenia on ≥2 occasions by end of study.
Time Frame: 6 months post transplant
Population: as for outcome 1
Measure: Number; unit: events
Arm/Group | Low Target Tacrolimus (Advagraf) | Standard Target Tacrolimus (Advagraf)
Number analyzed (Participants) | 14 | 14
events | 6 | 0

11. Secondary Outcome: Change From Baseline in Weight
Description: Any changes in weight by end of study.
Time Frame: baseline to 6 months post transplant
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: kg
Arm/Group | Low Target Tacrolimus (Advagraf) | Standard Target Tacrolimus (Advagraf)
Number analyzed (Participants) | 14 | 14
kg | 2.8 [0.8 to 6.8] | 1.5 [-1.3 to 3.8]

12. Secondary Outcome: eGFR at 6 Months
Description: Participant eGFR value by end of study.
Time Frame: 6 months post transplant
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: mL/min/1.73^2
Arm/Group | Low Target Tacrolimus (Advagraf) | Standard Target Tacrolimus (Advagraf)
Number analyzed (Participants) | 14 | 14
mL/min/1.73^2 | 56 [51 to 81] | 51 [43 to 63]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from the baseline visit until 6 months post transplant.
Arm/Group | Low Target Tacrolimus (Advagraf) | Standard Target Tacrolimus (Advagraf)
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 7/14 | 7/14
Other Adverse Events (participants affected / at risk) | 0/14 | 0/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Low Target Tacrolimus (Advagraf) (N=14) | Standard Target Tacrolimus (Advagraf) (N=14)
Dialysis (Renal and urinary disorders) | 2 | 2
Acute Rejection (Renal and urinary disorders) | 1 | 2
Malignancy (Immune system disorders) | 1 | 0
Infections (Infections and infestations) | 5 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-03): https://cdn.clinicaltrials.gov/large-docs/37/NCT01265537/Prot_SAP_000.pdf